CLINICAL TRIAL: NCT02892162
Title: Catheter Ablation Therapy for Persistent Atrial Fibrillation: Value of Additional Linear Ablation on Left Atrial Anterior Wall
Brief Title: Catheter Ablation Therapy for Persistent Atrial Fibrillation
Acronym: CLEAR-AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Beijing Hospital (Other Government); First Affiliated Hospital, Sun Yat-Sen University (Other); Tianjin Medical University General Hospital (Other); Wuhan Asia Heart Hospital (Other); First Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Principal Investigator, Yan Yao, MD,PhD, Principal Investigator, China National Center for Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-ZX51
Record Dates: First submitted 2016-08-27; First posted 2016-09-08 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Persistent Atrial Fibrillation
Keywords: atrial fibrillation; catheter ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- With additional LAAW linear ablation (Experimental): Patients who undergo CPVI+LA roof linear ablation+/ MI linear ablation, and additional LAAW linear ablation using ThermoCool SmartTouch catheter.
  Interventions: Procedure: Additional LAAW linear ablation
- Without additional LAAW linear ablation (Active Comparator): Patients who undergo CPVI+LA roof +/ MI linear ablation using ThermoCool SmartTouch catheter, without LAAW linear ablation.
  Interventions: Procedure: Additional LAAW linear ablation

INTERVENTIONS:
Procedure: Additional LAAW linear ablation — Additional linear ablation on LAAW using ThermoCool SmartTouch ablation catheter.

SUMMARY:
Use of catheter ablation for persistent atrial fibrillation (PerAF) remains controversial due to unsatisfactory long-term success rates (15% - 28.4%). The investigators' previous study indicated that the upper area of the left atrium (LA) plays an important role in PerAF, with the LA roof and mitral isthmus appearing to serve as main substrate in progression from PAF to PerAF and maintenance of fibrillatory activities. The investigators therefore hypothesized that AF should not be initiated or sustained if the latter crucial regions for AF maintenance are abolished. This study aimed to describe the efficacy and safety of additional linear ablation on the left atrial anterior wall for PerAF.

DETAILED DESCRIPTION:
Although studies and guidelines have helped establish catheter ablation as preferred treatment for patients suffering from paroxysmal atrial fibrillation (PAF), use of catheter ablation for persistent atrial fibrillation (PerAF) remains controversial due to unsatisfactory long-term success rates (15% - 28.4%).

The investigators' study indicated that the upper area of the left atrium (LA) plays an important role in PerAF, with the LA roof and mitral isthmus appearing to serve as main substrate in progression from PAF to PerAF and maintenance of fibrillatory activities. The investigators therefore hypothesized that AF should not be initiated or sustained if the latter crucial regions for AF maintenance are abolished. This was confirmed using a stepwise pure linear ablation protocol, consisting of a line across the LA roof and extending along the anterior wall of pulmonary veins (PV) antrum to mitral valve annulus (MVA) without PV isolation; the approach appeared safe and effective with long-term (5.2 years) follow-up success rate of 40% for PerAF.

This study will evaluate efficacy and safety of circumferential pulmonary vein isolation (CPVI) + LA roof linear ablation + LA anterior wall (LAAW) linear ablation combined with high density mapping and contact force sensing techniques for perAF. This study is expected to provide a practical and guided catheter ablation strategy with maximized safety and efficacy through use of contact force sensing technique, which will be accepted by other qualified electrophysiology laboratories.

ELIGIBILITY:
Inclusion Criteria:

- The main inclusion criterion is patients suffering from drug refractory persistent atrial fibrillation and referred to catheter ablation therapy. Persistent AF is defined as continuous AF for over 7 days, or lasting no more than 7 days but requiring pharmacological or electrical cardioversion.

Exclusion Criteria:

1. Patients without spontaneous ongoing AF at the beginning of the procedure;
2. Age: <18 years or >70 years;
3. LA size > 55mm measured on echocardiogram;
4. Previous AF ablation history including surgical ablation;
5. Documented LA thrombus;
6. Severe pulmonary diseases;
7. Previous cardiac surgical history.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
AF recurrence | From August, 2016 to July 2019. The overall Time Frame for AF recurrence is being assessed up to 36 months.
  Freedom from AF at 1 year without any anti-arrhythmic drugs. Recurrent AF is defined as documented AF (through 12-lead ECG or Holter) period lasting >30 seconds after a 3-month blanking period.

SECONDARY OUTCOMES:
Acute success rate of AF termination during ablation procedure | From August, 2016 to July 2017. The overall Time Frame for AF termination during ablation procedure is being assessed up to 12 months.
Frequency of complications | From August, 2016 to July 2017. The overall Time Frame for frequency of complications is being assessed up to 12 months.
Average radiation exposure | From August, 2016 to July 2017. The overall Time Frame for average radiation exposure is being assessed up to 12 months.
Frequency of redo procedures | From August, 2016 to July 2019. The overall Time Frame for frequency of redo procedures is being assessed up to 12 months.

OTHER OUTCOMES:
Average ablation time and procedure time | From August, 2016 to July 2017. The overall Time Frame for average ablation time and procedure time are being assessed up to 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Yao, MD,PhD, Principal Investigator — China National Center for Cardiovascular Diseases
Locations (1):
- China National Center for Cardiovascular Diseases, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; ACC/AHA Task Force Members. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: executive summary: a report of the American College of Cardiology/American Heart Association Task Force on practice guidelines and the Heart Rhythm Society. Circulation. 2014 Dec 2;130(23):2071-104. doi: 10.1161/CIR.0000000000000040. Epub 2014 Mar 28. No abstract available. PMID 24682348
- [Background] Camm AJ, Lip GY, De Caterina R, Savelieva I, Atar D, Hohnloser SH, Hindricks G, Kirchhof P; ESC Committee for Practice Guidelines (CPG). 2012 focused update of the ESC Guidelines for the management of atrial fibrillation: an update of the 2010 ESC Guidelines for the management of atrial fibrillation. Developed with the special contribution of the European Heart Rhythm Association. Eur Heart J. 2012 Nov;33(21):2719-47. doi: 10.1093/eurheartj/ehs253. Epub 2012 Aug 24. No abstract available. PMID 22922413
- [Background] Chao TF, Tsao HM, Lin YJ, Tsai CF, Lin WS, Chang SL, Lo LW, Hu YF, Tuan TC, Suenari K, Li CH, Hartono B, Chang HY, Ambrose K, Wu TJ, Chen SA. Clinical outcome of catheter ablation in patients with nonparoxysmal atrial fibrillation: results of 3-year follow-up. Circ Arrhythm Electrophysiol. 2012 Jun 1;5(3):514-20. doi: 10.1161/CIRCEP.111.968032. Epub 2012 May 1. PMID 22550126
- [Background] Tilz RR, Rillig A, Thum AM, Arya A, Wohlmuth P, Metzner A, Mathew S, Yoshiga Y, Wissner E, Kuck KH, Ouyang F. Catheter ablation of long-standing persistent atrial fibrillation: 5-year outcomes of the Hamburg Sequential Ablation Strategy. J Am Coll Cardiol. 2012 Nov 6;60(19):1921-9. doi: 10.1016/j.jacc.2012.04.060. Epub 2012 Oct 10. PMID 23062545
- [Background] Sorgente A, Tung P, Wylie J, Josephson ME. Six year follow-up after catheter ablation of atrial fibrillation: a palliation more than a true cure. Am J Cardiol. 2012 Apr 15;109(8):1179-86. doi: 10.1016/j.amjcard.2011.11.058. Epub 2012 Jan 14. PMID 22245414
- [Background] Yao Y, Zheng L, Zhang S, He DS, Zhang K, Tang M, Chen K, Pu J, Wang F, Chen X. Stepwise linear approach to catheter ablation of atrial fibrillation. Heart Rhythm. 2007 Dec;4(12):1497-504. doi: 10.1016/j.hrthm.2007.07.028. Epub 2007 Aug 11. PMID 17997359
- [Background] Wu L, Yao Y, Zheng L, Zhang K, Zhang S. Long-term follow-up of pure linear ablation for persistent atrial fibrillation without circumferential pulmonary vein isolation. J Cardiovasc Electrophysiol. 2014 May;25(5):471-476. doi: 10.1111/jce.12360. Epub 2014 Jan 24. PMID 24400694